CLINICAL TRIAL: NCT04124354
Title: Influence of Exercise on the Gut Microbiome of Overweight and Obese Adults With Prediabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 4 participants completed due to COVID-19 and the many lockdowns. We received a NIH R21 to complete a larger version of this trial and are working on launching this larger trial and submitting it to ClinicalTrials.gov.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00007532
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Experimental Group (Experimental): Participants will immediately begin an experimental supervised moderate-intensity treadmill walking intervention program.
  Interventions: Behavioral: Physical Activity
- Delayed Intervention Control Group (No Intervention): Participants will be asked to maintain their usual physical activity during the initial 8-week intervention period but will undergo all data collection procedures. Following the initial intervention period, these participants will be given the option to complete the 8-week intervention, with identical data collection procedures employed.

INTERVENTIONS:
Behavioral: Physical Activity — Participants will attend 3 treadmill walking sessions/week for 8 weeks (24 total)-exercising at 60-75% of their heart rate (HR) reserve monitored using Polar FT1 HR monitors. All walking sessions will take place using treadmills within the West Bank Office Building on the UMN-Twin Cities campus. Each walking session will be 30 min long during intervention weeks 1-4 and 45 min each during weeks 5-8. This exercise dose is equivalent to that employed in the only two human studies of exercise and the gut microbiome in addition to the dosage observed necessary to yield meaningful cardiometabolic changes. After the 4th- and 8th-weeks of the intervention, participants in both study groups will again undergo outcome assessments
  Arms: Immediate Experimental Group

SUMMARY:
Purpose: The investigators propose a 20-participant randomized 2-arm parallel trial with a delayed-intervention control examining how 8 weeks of moderate-intensity walking exercise alters the gut microbiome, short chain fatty acid (SCFA)-producing taxa, and the cardiometabolic profile and body weight of individuals who are overweight or obese and have prediabetes (PreD).

Aim 1: Examine and compare exercise-related shifts in the gut microbiome of individuals with PreD.

Aim 2: Examine and compare exercise-related changes in SCFA-producing taxa.

Exploratory Aim: Examine what percentage of the exercise-related changes observed in participants' gut microbiome and SCFA-producing taxa mediate changes in their cardiometabolic profile and body weight.

DETAILED DESCRIPTION:
In the U.S, 91.8 million adults have PreD. Preventing progression of PreD to type 2 diabetes (T2D) is vital. Odds of cardiovascular disease are higher among those with T2D, with $327 billion/year spent treating T2D. Major scientific organizations have thus called for studies of novel intermediates connecting health behaviors to pre-clinical cardiometabolic disease (CMD; e.g., PreD) to lower future clinical disease risk. Physical activity (PA) is key modifiable determinant of good health. PA recommendation adherence is associated with a 25-35% dose-dependent reduction in all-cause mortality, with as little as 75 min/week of regular moderate-intensity PA beneficial. In fact, an intervention within the Diabetes Prevention Program emphasizing PA participation at recommended levels was as successful as Metformin in preventing incident T2D-likely partially due to a 5kg-reduction in body weight during this trial. Yet, PA's impact on disease risk reduction is not explained entirely by CMD risk factors or weight loss, with mechanistic pathways still unclear and crucial to examine. The gut microbiota and microbiome have been posited as mechanistic intermediates linking PA to attenuated CMD development. However, there is no known research which has examined exercise-related changes in the human gut microbiome or SCFA-producing taxa in a population with a pre-clinical CMD such as PreD and how these changes mediate changes in CMD indices and body weight.

The proposed project is therefore innovative for a least two reasons. First, as stated, the investigators know of no study in individuals with PreD which examined how a moderate-intensity walking program may modify the gut microbiome and SCFA-producing taxa. Second, the investigators will use formal mediation analyses to examine the degree to which exercise-related changes in the gut microbiome and SCFA-producing taxa explain changes observed in CMD indices and body weight. These exploratory analyses will allow for a deeper interpretation of the physiological mechanisms by which exercise may improve health and inform future trial construction. Indeed, this study will provide critical preliminary evidence for a larger NIH R01-funded trial submitted to the NIDDK, NHLBI, or NCI, with the NIH committed to funding innovative scientific proposals involving the microbiome. The investigators will use this trial's observations to determine: 1) which taxa within the gut microbiome are most impacted by moderate-intensity walking; 2) the intra- and inter-person variability of gut microbiota changes due to moderate-intensity walking; and 3) whether the fixed frequency, intensity, and duration of the walking implemented results in meaningful changes. Observations in relation to these points will inform the design and implementation of future interventions to reduce pre-clinical disease states like PreD in a mechanistically-informed manner.

ELIGIBILITY:
Inclusion Criteria:

* Classified as overweight or obese with BMI 25.0-39.9 kg/m2
* Diagnosis of prediabetes as classified by a fasted blood glucose of 100 - 125 mg/dL, 2-hour oral glucose tolerance test of 140 - 199 mg/dL, or HbA1C level of 5.7% - 6.5%
* Currently engaged in < 150 minutes/week of physical activity-confirmed via the Modifiable Activity Questionnaire

Exclusion Criteria:

* Individuals with contraindications to exercise participation as assessed by the Physical Activity Readiness Questionnaire
* Self-reported physical/mental disabilities or gastrointestinal conditions
* Antibiotic usage within the last 45 days

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Shannon Index (Alpha-Diversity) as Reflected in Change in Operational Taxonomic Units | Baseline, 8 weeks
  Alpha diversity is the mean species diversity of a local site, which, in this study, is the fecal sample provided by participants used as a proxy for sampling the gut microbiome. The Shannon Index is based on the weighted geometric mean of the proportional abundances of the types of microbes. Change in alpha diversity will be reported as change in operational taxonomic units (OTUs).

SECONDARY OUTCOMES:
Change in Plasma LDL Concentrations | Baseline, 8 weeks
  Participants will have blood drawn after fasting over night or for at least 8 hours. Plasma low density lipoprotein (LDL) concentrations will be determined using standard laboratory assay methods. Concentrations will be reported in mg/dl.
Change in Plasma HDL Concentrations | Baseline, 8 weeks
  Participants will have blood drawn after fasting over night or for at least 8 hours. Plasma high density lipoprotein (HDL) concentrations will be determined using standard laboratory assay methods. Concentrations will be reported in mg/dl.
Change in Plasma Total Cholesterol Concentrations | Baseline, 8 weeks
  Participants will have blood drawn after fasting over night or for at least 8 hours. Plasma total cholesterol concentrations will be determined using standard laboratory assay methods. Concentrations will be reported in mg/dl.
Change in Plasma Insulin Concentrations | Baseline, 8 weeks
  Participants will have blood drawn after fasting over night or for at least 8 hours. Plasma insulin concentrations will be determined using standard laboratory assay methods. Concentrations will be reported in mmol/l.
Change in Plasma Glucose Concentrations | Baseline, 8 weeks
  Participants will have blood drawn after fasting over night or for at least 8 hours. Plasma glucose concentrations will be determined using standard laboratory assay methods. Concentrations will be reported in mg/dl.
Change in Plasma CRP Concentrations | Baseline, 8 weeks
  Participants will have blood drawn after fasting over night or for at least 8 hours. Plasma C-reactive protein (CRP) concentrations will be determined using standard laboratory assay methods. Concentrations will be reported in mg/l.
Change in Resting Blood Pressure - Systolic | Baseline, 8 weeks
  Resting blood pressure will be measured using an Omron Automatic BP Cuff and reported in mmHG.
Change in Resting Blood Pressure - Diastolic | Baseline, 8 weeks
  Resting blood pressure will be measured using an Omron Automatic BP Cuff and reported in mmHG.
Change in Waist Circumference | Baseline, 8 weeks
  Waist circumference will be measured using anthropometric tape and reported in cm.
Change in Body Weight | Baseline, 8 weeks
  Body weight will be measured using a Tanita Body Composition and Weight scale and reported in kg.
Change in Body Fat Percentage | Baseline, 8 weeks
  Body fat percentage will be measured using a Tanita Body Composition and Weight scale and reported as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Epidemiology Clinical Research Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No